CLINICAL TRIAL: NCT04288960
Title: Validity of a Belt Mounted Accelerometer to Assess Walking Measures in Patients With Chronic Stroke
Status: Suspended | Type: Observational
Why Stopped: Covid and access to participants
Sponsor: University of Winchester (Other)
Responsible Party: Sponsor
Other Study IDs: Wright_Validity_GWalk
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2021-11

CONDITIONS: Stroke; Gait, Hemiplegic
Keywords: stroke; validity; gait
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Stroke: Twenty chronic stroke patients (>3months post-stroke) will complete a one off session in a biomechanics lab. This session will include the Fugl Meyer Questionnaire and several walking trials along a flat, level 10m walkway. During this participants will wear a belt mounted accelerometer and small reflective markers on joints.
  Interventions: Device: Gwalk accelerometer walking trials

INTERVENTIONS:
Device: Gwalk accelerometer walking trials — No intervention. Participants will wear a belt mounted accelerometer and complete walking trials to assess validity of the device

SUMMARY:
The aim of this study is to validate the G-walk for several gait parameters, tested against a gold standard three dimensional camera system. This research will inform researchers and practitioners as to whether the G-Walk is a suitable and valid tool to easily assess walking ability in people with chronic stroke.

DETAILED DESCRIPTION:
Twenty chronic stroke survivors will be recruited for this study from an independent neuro-physiotherapy practice and community exercise programme.Gait analysis will be used to look at several gait parameters through the use of a three-dimensional visual analysis system based in our Biomechanics Lab at the University of Winchester. Participants will attend testing one testing session of approximately 1 hour. During this testing session functional measures and walking trials will be assessed. Participants will first be asked to complete a set of simple movements that will contribute towards Fugl Meyer questionnaire. Twenty eight reflective markers will then be attached to specified joints and segments of the body, such as the thigh, with double sided sticky tape to allow for data collection through the camera system to collect kinematic data. The belt mounted accelerometer (G-Walk) will be positioned around the waist over the L5 vertebrae. Participants will be asked to perform 6 walking trials of 10m to collect 3D kinematic and accelerometer gait data.

ELIGIBILITY:
Inclusion Criteria:

* <3 months post stroke
* Lower limb impairment
* Able to stand and step independently
* Functional ambulation classifications (FAC) of 2-5
* Modified Rankin Scale (MRS) of 1-3
* Cognitively aware to undertake the testing session

Exclusion Criteria:

* Unresolved deep vein thrombosis
* unstable cardiovascular conditions
* open wounds
* active drug resistant infection
* recent fractures of involved limb
* peripheral arterial disease
* incontinence
* severe osteoporosis
* non-weight bearing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic stroke (<3month post stroke) will be recruited from a neuro-physiotherapy practice, community-based stroke support groups and community exercise programme. All participants would have been diagnosed with stroke by a specialist neurologist/stroke consultant from a UK National Health Service (NHS) Foundation Trust, and have undertaken normal inpatient and outpatient rehabilitation in accordance with NICE guidelines (National Institute of Health and CARE
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Speed | 60 minutes
  How quickly a participant walks overground
Cadence | 60 minutes
  Steps taken per minute
Stride Length | 60 minutes
  The distance between strides
Swing phase duration | 60 minutes
  Percentage of the gait cycle spent in swing phase
Stance phase duration | 60 minutes
  Percentage of the gait cycle spent in stance phase
Gait cycle duration | 60 minutes
  The time it takes to complete one gait cycle
Double support duration | 60 minutes
  Percentage of the gait cycle spend with both feet on the ground (double support)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Wright, MSc, Principal Investigator — University of Winchester
Locations (1):
- University of Winchester, Winchester, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share this information with other researchers

REFERENCES:
- [Background] De Ridder R, Lebleu J, Willems T, De Blaiser C, Detrembleur C, Roosen P. Concurrent Validity of a Commercial Wireless Trunk Triaxial Accelerometer System for Gait Analysis. J Sport Rehabil. 2019 Aug 1;28(6):jsr.2018-0295. doi: 10.1123/jsr.2018-0295. PMID 30747572